

#### **Informed Consent**

# INFORMED CONSENT/AUTHORIZATION FOR PARTICIPATION IN RESEARCH

A Phase I-II Study Investigating the All Oral Combination of the Menin Inhibitor SNDX-5613 with Decitabine/Cedazuridine (ASTX727) and Venetoclax in Acute Myeloid Leukemia (SAVE-ML)

2021-1059

| Subtitle: Protocol V.05, January 28, 2025 | 5 | |
|-------------------------------------------|-----------------------|---|
| Study Chair: Ghayas Issa | | |
| Participant's Name | Medical Record Number | - |

This is an informed consent and authorization form for a research study. It includes a summary about the study. A more detailed description of procedures and risks is provided after the summary.

This research has been reviewed and approved by an Institutional Review Board (IRB - a committee that reviews research studies).

If you are reading and signing this form on behalf of a potential participant, please note: Any time the words "you," "your," "I," or "me" appear, it is meant to apply to the potential participant.

#### STUDY SUMMARY

There are 2 parts to this study: Part 1b (dose escalation) and Part 2 (dose expansion).

The goal of Part 1b of this clinical research study is to find the highest tolerable dose of revumenib (SNDX-5613) that can be given in combination with ASTX727 (a combination of the drugs decitabine/cedazuridine) and venetoclax for patients with acute myeloid leukemia (AML) or those with a mixed phenotype acute leukemia with a myeloid phenotype (MPAL).

The goal of Part 2 of this study is to learn if the dose of study drugs found in Part 1b can help to control AML/MPAL that is newly diagnosed, relapsed (has come back after treatment), or refractory (is resistant to treatment).

The safety of these study drug combinations will also be studied.

This is an investigational study. SNDX-5613 is not FDA approved or commercially available. It is currently being used for research purposes only. ASTX727 is FDA approved and commercially available for the treatment of myelodysplastic syndromes (MDS). Venetoclax is FDA approved and commercially available for the treatment of AML and chronic lymphocytic leukemia/small lymphocytic lymphoma (CLL/SLL). The treatment combinations that are given in this study are considered investigational.

The study drugs may help to control the disease. Future patients may benefit from what is learned. There may be no benefits for you in this study.

Your participation is completely voluntary. Before choosing to take part in this study, you should discuss with the study team any concerns you may have, including side effects, potential expenses, and time commitment.

You can read a list of potential side effects below in the Possible Risks section of this consent.

Your participation in this study may last up to about 3 years, depending on how you tolerate the study drugs.

SNDX-5613 and ASTX727 will be provided at no cost to you during the study. You and/or your insurance provider will be responsible for the cost of all other treatment given on study.

You may choose not to take part in this study. Instead of taking part in the study, you may choose to receive other standard, FDA-approved therapy. There are many treatment options for leukemia. The study doctor will talk to you about which treatment options may be available outside of this study, including their possible risks and benefits. You may choose to receive other investigational therapy, if available. You may choose not to have treatment for cancer at all. In all cases, you will receive appropriate medical care, including treatment for pain and other symptoms of cancer.

#### 1. STUDY DETAILS

#### **Screening Tests**

Signing this consent form does not mean that you will be able to take part in this study. The following screening tests will help the doctor decide if you are eligible:

- You will have a physical exam.
- You will have an eye exam to check your eye health and your vision. If this is not done at screening, it may be done within 7 days after your first dose of SNDX-5613.
- You will have a triplicate EKG (3 EKGs in a row) and either an echocardiogram (ECHO) or MUGA scan to check your heart function.

- Blood (about 2 teaspoons) will be drawn for routine tests.
- You will have a bone marrow biopsy/aspirate to check the status of the disease, for research testing, and for cytogenetic testing. Cytogenetic testing looks at how genetic changes to cells may affect how the disease may react to the study drug. In this study, research testing refers to special types of tests done to understand how or why your body responds (or does not respond) to the study treatments. To collect a bone marrow biopsy/aspirate, an area of the hip or other site is numbed with anesthetic, and a small amount of bone marrow and bone is withdrawn through a large needle.
- If you can become pregnant, urine or blood (about 1 teaspoon) will be collected for a pregnancy test. To take part in this study, you must not be pregnant.

The study doctor will discuss the screening test results with you. If the screening tests show that you are not eligible to take part in the study, you will not be enrolled. Other treatment options will be discussed with you.

#### **Study Groups**

If you are found to be eligible to take part in this study, you will be assigned to a study group based on when you join this study. Up to 12 participants will be enrolled in Phase I of the study, and up to 54 participants total will be enrolled in both cohorts of Phase II.

If you are enrolled in **Phase I**, the dose of SNDX-5613 you receive will depend on when you join this study and whether or not you are taking a type of drug called a CYP3A4 inhibitor. The first group of participants will receive the starting dose level(s) of SNDX-5613. The next dosing group will receive a higher dose of SNDX-5613 than the group before it, if no intolerable side effects were seen. If intolerable side effects are seen, a dose level lower than the starting dose will be tested with the second dosing group.

At each assigned dose level, participants who are not also taking a CYP3A4 inhibitor will receive a higher dose level than others in their dosing group who are taking CYP3A4 inhibitor drugs.

If you are enrolled in **Phase II**, you will receive SNDX-5613 at the recommended dose that was found in Phase I.

Your dose of venetoclax and ASTX727 will not change.

Up to 66 participants will be enrolled in this study. All will take part at MD Anderson.

#### **Study Drug Administration**

Each study cycle is 28 days.

You will take **SNDX-5613** capsules or tablets by mouth 2 times every day (about 12 hours apart). The exact dose or dosing interval may be adjusted throughout your

treatment. You should take the drug on an empty stomach (at least 1 hour before or 2 hours after a meal). However, you may take SNDX-5613 with a low-fat meal on days when you do not receive ASTX727. The capsules/tablets should be swallowed whole with about 1 cup of water.

If you cannot swallow capsules whole, a liquid formulation may be taken by mouth or given through a nasogastric or gastrostomy tube (special tube that carries food and medicine to the stomach through the nose or abdomen). Your doctor can discuss these options with you, if needed.

SNDX-5613 capsules or its liquid formulation must be stored in the refrigerator in their original container. Do not transfer capsules to a pill case or other container. You must bring back any empty bottles or leftover capsules in their original container to your next clinic visit.

#### You will also take:

- Venetoclax tablets by mouth on Days 1-14 of each cycle.
  - Venetoclax must be taken with at least 8 ounces (1 cup) of water within 30 minutes after eating, preferably a low or moderate-fat breakfast.
  - Do not have grapefruit or grapefruit-containing products, Seville (sour) oranges, or star fruit while taking venetoclax.
  - If you miss a dose, you may make up the dose later in the day as long as it is within 6 hours after the missed dose. If more than 6 hours have passed, skip that dose and take your next dose as scheduled.
  - If you vomit a dose, do not make it up. Wait and take your next dose as scheduled.
- ASTX727 tablets by mouth on Days 1-5 of each cycle.
  - ASTX727 must be taken on an empty stomach (no food or water for 2 hours before and after meals). Tablets should be taken whole; do not chew or crush them.
  - If you miss a dose, take it as soon as possible (as long as it is within 12 hours of the missed dose time). If more than 12 hours have passed, skip that dose and take your next dose as scheduled.
  - If you vomit a dose, do not make it up. Wait and take your next dose as scheduled.
  - Contact the study doctor right away if any of the tablets you receive are broken. You should not take or touch broken tablets. You will be given replacement tablets.

You may be given cytarabine or methotrexate directly into the spinal fluid (called intrathecal chemotherapy) if leukemia cells are found in the spinal fluid or if you are at high-risk of developing leukemia in the spinal fluid and the brain in the future. You will sign a separate consent for this procedure which explains the procedure and its risks in detail.

You will be given standard drugs to help decrease the risk of side effects. You may ask the study staff for information about how the drugs are given and their risks.

You may also begin taking a type of anti-fungal medication (called a strong CYP3A4 inhibitor) for at least 7 days before your first dose of study drug(s) and while receiving SNDX-5613. This may depend on what standard treatments are recommended, your health status, past treatments, insurance limitations, and other factors. You will not be able to receive any other type of this medication. The study doctor will discuss which anti-fungal medication you will receive and how to take them. Examples of medications you may be given include:

- Itraconazole
- Ketoconazole
- Posaconazole
- Voriconazole

You will be given a study drug diary to write down when you take each dose of SNDX-5613 and your other assigned doses (if they are taken by mouth at home). You should write down if you miss or vomit any doses. Bring your drug diary and your medications with you to each clinic visit.

You will no longer be able to take the study drugs if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

#### **Study Visits**

## On Days 1, 8, 14, and 22 of Cycles 1 and 2:

- Blood (about 2 teaspoons) will be drawn for routine tests. On Day 1 of Cycle 1, blood (about 2 tablespoons) will also be drawn for research testing. If you are receiving venetoclax, part of this blood sample will be used to check for signs of tumor lysis syndrome (TLS), a side effect of venetoclax. This is described in more detail below under "Possible Risks."
- If you are in Phase I only, blood (about 1/2 teaspoon each time) will be drawn for pharmacokinetic (PK) testing on Days 8 and 15 of Cycle 1 and Day 1 of Cycle 2. PK testing measures the amount of study drug in the body at different time points.
- In Cycle 1 only, you will have a triplicate EKG before the dose and then at 2 hours after the dose. If the study doctor thinks it is needed, you may have another triplicate EKG at 4 hours after the dose.
- On Day 1 only:
  - You will have a physical exam.
  - Starting at Cycle 4 and every 3 cycles after that (Cycles 7, 10, 13, and so on), as long as the doctor thinks it is needed, you will have an eye exam to check your eye health and your vision.
  - If you can become pregnant, urine or blood will be collected for a pregnancy test (Cycle 1 only).

#### On Days 2-4 of Cycle 1:

Blood (about 2 teaspoons) will be drawn to check for signs of TLS.

 On Day 3 only, you will have a triplicate EKG before the dose and then at 2 hours after the dose. If the study doctor thinks it is needed, you may have another triplicate EKG at 4 hours after the dose.

On **Day 14 of Cycle 1**, you may have a bone marrow aspirate/biopsy to check the status of the disease. Depending on the results of that biopsy, you may be told to stop taking SNDX-5613, starting on Day 21. The study team can discuss this with you further.

On **Day 5 of Cycle 2**, you will have a triplicate EKG before the dose and then at 2 hours after the dose. If the study doctor thinks it is needed, you may have another triplicate EKG at 4 hours after the dose.

## Between Days 21 and 28 of Cycles 1, 3, 5, and every 3 cycles after that (Cycles 8, 11, 13, and so on):

- You will have a bone marrow biopsy/aspirate to check the status of the disease and for research testing.
- Blood (about 2 tablespoons) will be drawn for research testing (Cycles 1, 3, and 5 only).

If the disease appears to get worse, you will have a bone marrow biopsy/aspirate and blood drawn for research testing.

## On Day 1 of Cycles 3 and beyond:

- You will have a physical exam.
- Blood (about 2 ½ teaspoons) will be drawn for routine tests. If you are receiving venetoclax, part of this blood sample will be used to check for signs of TLS.
- You will have a triplicate EKG. In Cycle 3 only, you will have triplicate EKG before the dose and then at 2 hours after the dose. If the study doctor thinks it is needed, you may have another triplicate EKG at 4 hours after the dose.
- If you are in Phase I, on Day 1 of Cycle 3 only, blood (about 1/2 teaspoon each time) will be drawn for PK tests.

#### **End-of-Dosing Visit**

Within 30 days after your last dose of study drugs:

- You will have a physical exam.
- Blood (about 2½ tablespoons) will be drawn for routine tests and research testing.
- If one has not been done in the last month, you will have an eye exam.
- If the doctor thinks it is needed, you may have a bone marrow biopsy/aspirate.

## **Follow-Up Visits**

Every month for up to 3 years after the last participant has enrolled in the study, the study team will call you and ask how you are doing and if you have started any new anti-cancer medications. Each call should last about 5-10 minutes.

#### Other Information

While in this study, you should avoid certain medications and foods (like grapefruit and grapefruit juice). It is important to tell the study doctor about all medications you are taking or plan to take (including prescription and over-the-counter medications, herbal remedies, vitamins, and/or supplements).

The study doctor will tell you which medications and foods you should avoid during the study.

#### 2. POSSIBLE RISKS

While on this study, you are at risk for side effects. You should discuss these with the study doctor. The more commonly occurring side effects are listed in this form, as are rare but serious side effects. You may also want to ask about uncommon side effects that have been observed in small numbers of patients but are not listed in this form. Many side effects go away shortly after treatment is stopped, but in some cases side effects may be serious, long-lasting or permanent, and may even result in hospitalization and/or death.

Side effects will vary from person to person, and some may occur after you have stopped receiving treatment. Tell the study staff about any side effects you may have, even if you do not think they are related to the study drugs/procedures.

SNDX-5613, venetoclax, ASTX727, itraconazole, ketoconazole, posaconazole, and voriconazole may cause a low blood cell count (red, platelets, and/or white blood cells):

- A low red blood cell count (anemia) may cause difficulty breathing and/or fatigue. You may need a blood transfusion.
- A low platelet count increases your risk of bleeding (such as nosebleeds, bruising, stroke, and/or digestive system bleeding). You may need a platelet transfusion.
- A low white blood cell count increases your risk of infection (such as pneumonia and/or severe blood infection). Infections may occur anywhere and become life-threatening. Symptoms of infection may include fever, pain, redness, and difficulty breathing.

## **SNDX-5613 Side Effects**

This is an early study of SDX-5613 in humans, so the side effects are not well known. Based on studies in animals, SDX05613 may cause the following side effects:

| abnormal EKG | increased size of | problems with |
|---------------------|---------------------------|------------------------|
| increased size of | pituitary gland (possible | production of sperm or |
| thyroid/parathyroid | vision problems or | eggs |
| | headaches) | |

| glands (possible goiter<br>[mass] in the neck) | <ul> <li>enlarged mammary glands</li> <li>death of prostate tissue (possible overactive bladder)</li> </ul> | <ul> <li>abnormal liver test (possible liver damage)</li> <li>fatty liver (possible liver damage)</li> <li>cataracts (clouding of the lens of the eye)</li> <li>nausea</li> <li>vomiting</li> </ul> |
|---|---|---|
|---|---|---|

SNDX-5613 may cause you to develop differentiation syndrome (sometimes called retinoic acid syndrome). Differentiation syndrome is a serious or possibly life-threatening condition that may cause possible increase in the white blood cell count, fever, difficulty breathing, swelling, altered mental status and/or kidney failure. Call your healthcare provider or go to the nearest hospital emergency room right away if you develop any of the following symptoms of differentiation syndrome during treatment with SNDX-5613:

- fever
- cough
- trouble breathing
- skin rash
- decreased urination
- dizziness or lightheadedness
- rapid weight gain
- swelling of your arms or legs

If you develop signs and symptoms of differentiation syndrome, your healthcare provider may treat you with a corticosteroid medicine or a medicine called hydroxyurea and may monitor you in the hospital.

SNDX-5613 may affect the electricity of the heart manifesting as a change in the EKG pattern called QT prolongation which may lead to life-threatening changes in the heart rhythm. Very low potassium or magnesium blood levels increase this risk and therefore should be corrected using potassium or magnesium supplementation while taking SNDX-5613.

Patients receiving strong CYP3A4 inhibitors such as itraconazole, ketoconazole, posaconazole, or voriconazole may have an increased risk of these side effects as it may take the body longer to clear SNDX-5613 from their blood.

## **Venetoclax Side Effects**

## Common (occurring in more than 20% of patients)

| swelling (arm/leg) | <ul><li>diarrhea</li></ul> | muscle and/or bone |
|--------------------|----------------------------|--------------------|
| fatigue | <ul><li>nausea</li></ul> | pain |

- high blood sugar (possible diabetes)
- abnormal salts,
   minerals, and/or acids
   in the blood (possible
   weakness, swelling,
   fatigue, low blood
   pressure, organ failure,
   heart problems,
   changes in mental
   status, and/or seizure)
- low blood counts (red, platelets, and white)
- abnormal liver tests (possible liver damage)
- upper respiratory tract infection
- cough

## Occasional (occurring in 3-20% of patients)

- fever
- headache
- dizziness
- skin rash
- vomiting
- constipation
- abdominal pain
- mouth blisters/sores (possible difficulty swallowing)
- joint pain

- high blood levels of uric acid (possible painful joints and/or kidney failure)
- pneumonia
- difficulty breathing
- severe life-threatening infection (possible low blood pressure, kidney failure, and/or heart failure)
- bacteria in the blood
- tumor lysis syndrome (TLS)--breakdown products of the cancer cells entering the blood stream (possible weakness, low blood pressure, muscle cramps, kidney damage, and/or other organ damage)

TLS is a problem that can occur when cancer cells break down rapidly and the body has to get rid of the broken up cell parts. Sometimes your body, especially the kidneys, cannot remove the cell parts quickly enough, so the level of some of these cell products in your blood, such as salts and acids, can rise. This can happen especially in participants with large tumors or a high number of cancerous white cells in the blood. TLS can lead to serious problems, such as effects on your kidneys and heart (including abnormal heart rhythms), seizures, or even death.

If you develop TLS, your urine may look dark, thick, or cloudy. You may have fever, chills, nausea/vomiting, diarrhea, confusion, shortness of breath, irregular heartbeat, fatigue, muscle pain, joint discomfort, and/or seizure. If you notice any of these, tell your doctor or nurse right away. Your study doctor will closely watch and treat you as needed to lower the risk of any serious changes in your blood or other complications of TLS. You may need to have extra blood tests or EKGs to check for signs of TLS.

You should wear ear plugs or other hearing protection when involved in a loud activity.

If you notice any rash, hives, itching, or other signs of an allergic reaction such as swelling, wheezing, or you are having a hard time breathing, tell your doctor right away.

At this time, there are no known serious side effects that occur in fewer than 3% of patients.

## **ASTX727 Side Effects**

## Common (occurring in more than 20% of patients)

| <ul> <li>fatigue</li> <li>headache</li> <li>low blood level of<br/>albumin (possible<br/>swelling, weakness,</li> </ul> | <ul><li>nausea</li><li>low blood cell counts<br/>(red, white, platelets)</li></ul> | abnormal liver tests (possible liver damage) |
|---|---|---|
| and/or fatigue) | | |

If you experience fever or other signs and symptoms of infection or bleeding, you should contact your study doctor or study nurse right away and seek medical attention.

## Occasional (occurring in 3-20% of patients)

| <ul> <li>irregular heartbeat</li> <li>swelling</li> <li>low blood pressure (possible dizziness and/or fainting)</li> <li>falls</li> <li>fever</li> <li>difficulty sleeping</li> <li>nerve damage (loss of motor or sensory function)</li> <li>dizziness</li> <li>skin rash</li> <li>low blood sugar (possible diabetes)</li> </ul> | <ul> <li>low blood levels of calcium (possible weakness and/or cramping)</li> <li>low blood levels of sodium (possible headache, confusion, seizures, and/or coma)</li> <li>constipation</li> <li>diarrhea</li> <li>weight loss</li> <li>abdominal pain</li> <li>loss of appetite</li> <li>vomiting</li> <li>heartburn (acid reflux)</li> </ul> | <ul> <li>mouth blisters/sores (possible difficulty swallowing)</li> <li>joint/muscle pain</li> <li>abnormal kidney test (possible kidney damage)</li> <li>decreased kidney function</li> <li>difficulty breathing</li> <li>cough</li> </ul> |
|---|---|---|

## Rare but serious (occurring in fewer than 3% of patients)

| bleeding in the brain | <ul> <li>lung inflammation</li> </ul> | tumor lysis syndrome |
|---|---|---|
| <ul> <li>clubbing (changes in</li> </ul> | (possible difficulty | (TLS)breakdown |
| the areas around the | breathing) | products of the cancer |

| toenails/fingernails), | cells entering the blood |
|------------------------|--------------------------|
| which can be serious | stream (possible |
| | weakness, low blood |
| | pressure, muscle |
| | cramps, kidney |
| | damage, and/or other |
| | organ damage) |

In rare cases (may affect from 1 in 1000 people to 1 in 10,000 people), these reactions to ASTX727 have been reported:

- Hypersensitivity (allergic) reaction related to the drug, which could include one
  or more of the following: rash; hives; swelling of the face, lips, tongue, or
  throat; and difficulty swallowing or breathing.
- ASTX727 may cause Sweet's syndrome (acute neutrophilic dermatosis): a condition that may include cough, shortness of breath, fever, and a painful rash on the arms, legs, trunk, face, or neck.

The side effects from ASTX727 are expected to be similar to those from decitabine given by vein. Based on the decitabine risks, there is also a rare possibility that ASTX727 may cause differentiation syndrome or interstitial lung disease (described below). However, these events have not been reported in ASTX727 studies so far.

- Differentiation Syndrome may cause fever, cough, difficulty breathing, weight gain, swelling of the arms, legs, and/or neck, build-up of fluid around the heart and lungs, low blood pressure, and/or kidney failure.
- Interstitial lung disease: may include sudden shortness of breath, tiredness, dry cough, and generally feeling unwell. This can be a serious complication requiring treatment.

**Using the study drugs together** may cause side effects that are not seen when each is given alone. The study drug combination may also increase the frequency and/or severity of the side effects listed above.

#### Other Risks

**EKGs and ECHOs** may cause discomfort while lying on the exam table, and the tape on the EKG pads may cause skin irritation.

**MUGA scans** may cause allergic reactions to the radioactive tracer, injection site soreness, and/or swelling. They may cause damage to cells or tissue from being exposed to the radiation used in the scan. These side effects may occur in less than 10% of patients.

**Blood draws** may cause pain, bleeding, and/or bruising. You may faint and/or develop an infection with redness and irritation of the vein at the site where blood is drawn. Frequent blood collection may cause anemia (low red blood cell count), which may create a need for blood transfusions.

Having **bone marrow biopsies/aspirates** performed may cause pain, bruising, bleeding, redness, low blood pressure, swelling, and/or infection at the site of the biopsies/aspirates. An allergic reaction to the anesthetic may occur. A scar may form at the biopsy/aspirate site.

This study may involve unpredictable risks to the participants.

#### **Confidentiality Risk**

Although every effort will be made to keep study data safe, there is a chance that your personal health information could be lost or stolen, which may result in a **loss of confidentiality**. All study data will be stored in password-protected computers and/or locked file cabinets and will continue to be stored securely after the study.

#### **Pregnancy Related Risks**

Taking part in this study can result in risks to an unborn or breastfeeding baby, so you should not become pregnant, breastfeed a baby, or father a child while on this study.

If you can become pregnant or father a child, you must use birth control during the study and for at least 3 months after your last dose of study treatment, if you are sexually active.

Talk to the study doctor about acceptable methods of birth control to use during the study.

Males: Tell the doctor right away if your partner becomes pregnant or suspects pregnancy.

Females: If you are pregnant, you will not be enrolled on this study. If you become pregnant or suspect that you are pregnant, you must tell your doctor right away.

Getting pregnant will result in your removal from this study.

#### 3. COSTS AND COMPENSATION

If you suffer injury as a direct result of taking part in this study, MD Anderson health providers will provide medical care. However, this medical care will be billed to your insurance provider or you in the ordinary manner. You will not be reimbursed for expenses or compensated financially by MD Anderson, Taiho Oncology, or Syndax Pharmaceuticals for this injury. You may also contact the Chair of MD Anderson's IRB at 713-792-6477 with questions about study-related injuries. By signing this consent form, you are not giving up any of your legal rights.

Certain tests, procedures, and/or drugs that you may receive as part of this study may be without cost to you because they are for research purposes only. However, your insurance provider and/or you may be financially responsible for the cost of care and treatment of any complications resulting from the research tests,

procedures, and/or drugs. Standard medical care that you receive under this research study will be billed to your insurance provider and/or you in the ordinary manner. Before taking part in this study, you may ask about which parts of the research-related care may be provided without charge, which costs your insurance provider may pay for, and which costs may be your responsibility. You may ask that a financial counselor be made available to you to talk about the costs of this study.

Samples that are collected from you in this study may be used for the development of treatments, devices, new drugs, or patentable procedures that may result in commercial profit.

There are no plans to compensate you for any patents or discoveries that may result from your participation in this research.

You will receive no compensation for taking part in this study.

### **Additional Information**

- 4. You may ask the study chair (Dr. Ghayas Issa, at 713-745-6798) any questions you have about this study. You may also contact the Chair of MD Anderson's Institutional Review Board (IRB a committee that reviews research studies) at 713-792-6477 with any questions that have to do with this study or your rights as a study participant.
- 5. You may choose not to take part in this study without any penalty or loss of benefits to which you are otherwise entitled. You may also withdraw from participation in this study at any time without any penalty or loss of benefits. If you decide you want to stop taking part in the study, it is recommended for your safety that you first talk to your doctor who can help you safely stop study treatment. It may be dangerous to suddenly stop study treatment. The study doctor will also decide if you need to have any visits or tests to check on your health. If you withdraw from this study, you can still choose to be treated at MD Anderson.

If you stop being in the research, already collected data may not be removed from the study database. You may be asked whether the study doctor can collect data from your routine medical care. If you agree, this data will be handled the same as research data.

- 6. This study or your participation in it may be changed or stopped without your consent at any time by the study chair, Taiho Oncology, Syndax Pharmaceuticals, the U.S. Food and Drug Administration (FDA), the Office for Human Research Protections (OHRP), or the IRB of MD Anderson. Possible reasons your participation in this study may be stopped include if the disease gets worse, if intolerable side effects occur, if you are unable to follow study directions, or if the study is stopped.
- 7. You will be informed of any new findings or information that might affect your willingness to continue taking part in the study and you may be asked to sign

another informed consent and authorization form stating your continued willingness to participate in this study.

- 8. MD Anderson may benefit from your participation and/or what is learned in this study.
- 9. This study is sponsored and/or supported by: Taiho Oncology and Syndax Pharmaceuticals
- 10. In a medical emergency, you may be cared for by someone who has a financial interest with the study sponsor(s)/supporter. If you have any questions about this, you may call the IRB at 713-792-6477.

#### **Future Research**

#### Data

Your personal information is being collected as part of this study. These data may be used by researchers at MD Anderson, Taiho Oncology, Syndax Pharmaceuticals, and/or shared with other researchers and/or institutions for use in future research.

The study staff may ask if they can continue collecting the results of routine care from your medical record.

#### **Samples**

Samples (such as blood and/or tissue) are being collected from you as part of this study. Researchers at MD Anderson may use any leftover samples that are stored at MD Anderson in future research. Leftover samples will not be stored by Taiho Oncology or Syndax Pharmaceuticals used in future research.

Before being used or shared for future research, every effort will be made to remove your identifying information from any data and/or research samples. If all identifying information is removed, you will not be asked for additional permission before future research is performed.

In some cases, all of your identifying information may not be removed before your data or research samples are used for future research. If future research is performed at MD Anderson, the researchers must get approval from the Institutional Review Board (IRB) of MD Anderson before your data and/or research samples can be used. At that time, the IRB will decide whether or not further permission from you is required. The IRB is a committee of doctors, researchers, and community members that is responsible for protecting study participants and making sure all research is safe and ethical.

If this research is not performed at MD Anderson, MD Anderson will not have oversight of any data and/or samples.

#### **Genetic Research**

Research samples collected from you as part of this study may be used for genetic research, which may include whole genome sequencing. Whole genome sequencing is a type of testing in which researchers study your entire genetic makeup (DNA). This may help researchers learn how changes in the ordering of genes may affect a disease or response to treatment. If genetic research is done with your samples, those who have access to those samples may be able to identify you. The results of this research may also be able to be linked to you.

If genetic research is done with your samples, those who have access to those samples may be able to identify you. The results of this research may also be able to be linked to you. The same level of data protection that covers your individual data does not apply to summary results (when data from the whole study is combined).

A federal law, called the Genetic Information Nondiscrimination Act (GINA), generally makes it illegal for health insurance companies, group health plans, and most employers to discriminate against you based on your genetic information. This law generally will protect you in the following ways:

- Health insurance companies and group health plans may not request your genetic information that we get from this research.
- Health insurance companies and group health plans may not use your genetic information when making decisions regarding your eligibility or premiums.
- Employers with 15 or more employees may not use your genetic information that we get from this research when deciding to hire, promote, or fire you or when setting the terms of your employment.

Be aware that this federal law does not protect you against genetic discrimination by companies that sell life insurance, disability insurance, or long-term care insurance. Nor does this federal law prohibit discrimination based on an already known genetic disease or disorder.

## **Conflict of Interest**

Outside relationships are disclosed to and approved by the Conflict of Interest Committee, which reviews these relationships for compliance with institutional policy. This review helps the IRB to assure that financial relationships do not have an impact on the conduct of this study. The following members of the study staff have disclosed compensation from the funding source(s) of this study:

- Ghayas Issa (Principal Investigator)
- Tapan Kadia, Elias Jabbour, Naval Daver, and Branko Cuglievan (Co-Investigators)

## <u>Authorization for Use and Disclosure of Protected Health Information (PHI):</u>

A. During the course of this study, MD Anderson will be collecting and using your PHI, including identifying information, information from your medical record, and study results. For legal, ethical, research, and safety-related reasons, your doctor and the research team may share your PHI with:

- Federal agencies that require reporting of clinical study data (such as the FDA, National Cancer Institute [NCI], and OHRP)
- The IRB and officials of MD Anderson
- Taiho Oncology and Syndax Pharmaceuticals, who are sponsors or supporters of this study, and/or any future sponsors/supporters of the study
- Study monitors and auditors who verify the accuracy of the information
- Individuals who put all the study information together in report form

Study sponsors and/or supporters receive limited amounts of PHI. They may also view additional PHI in study records during the monitoring process. MD Anderson's contracts require sponsors/supporters to protect this information and limit how they may use it.

The results of this research may be published in scientific journals or presented at medical meetings, but your identity will not be disclosed.

- B. Signing this consent and authorization form is optional but you cannot take part in this study or receive study-related treatment if you do not agree and sign.
- C. MD Anderson will keep your PHI confidential when possible (according to state and federal law). However, in some situations, the FDA could be required to reveal the names of participants.

Once disclosed outside of MD Anderson, federal privacy laws may no longer protect your PHI.

D. The permission to use your PHI will continue indefinitely unless you withdraw your authorization in writing. Instructions on how to do this can be found in the MD Anderson Notice of Privacy Practices (NPP) or you may contact the Chief Privacy Officer at 713-745-6636. If you withdraw your authorization, you will be removed from the study and the data collected about you up to that point can be used and included in data analysis. However, no further information about you will be collected.

If you leave the study early (withdraw), you will be asked if the study team can collect information from your medical record about your routine medical care. This may help researchers better understand the long-term effects of the study drugs.

E. A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

Protocol 2021-1059 NCT05360160 January 28, 2025 

## CONSENT/AUTHORIZATION (Adult Participants Only)

I understand the information in this consent form. I have had a chance to read the consent form for this study, or have had it read to me. I have had a chance to think about it, ask questions, and talk about it with others as needed. I give the study chair permission to enroll me on this study. By signing this consent form, I am not giving up any of my legal rights. I will be given a signed copy of this consent document.

| SIGNATURE OF PARTICIPANT | DATE |
|---|---|
| PRINTED NAME OF PARTICIPANT | |
| WITNESS TO CONSENT | |
| I was present during the explanation of the research to be performed | under this protocol. |
| SIGNATURE OF WITNESS TO THE VERBAL CONSENT PRESENTATION (OTHER THAN PHYSICIAN OR STUDY CHAIR) | DATE |
| A witness signature is only required for non-English speakers utilizing the | |
| short form consent process (VTPS) and patients who are illiterate. | |
| PRINTED NAME OF WITNESS TO THE VERBAL CONSENT | |
| PERSON OBTAINING CONSENT | |
| I have discussed this research study with the participant and/or his o | r her authorized |
| representative, using language that is understandable and appropria | |
| have fully informed this participant of the nature of this study and its participant of the nature of th | possible benefits |
| and risks and that the participant understood this explanation. | |
| PERSON OBTAINING CONSENT | DATE |
| PRINTED NAME OF PERSON OBTAINING CONSENT | |

Protocol 2021-1059 NCT05360160 January 28, 2025 

## **PARENT/GUARDIAN PERMISSION**

| discuss the study and ask questions. My questions have been answer permission for my child or ward to take part in this study. | ed. I give |
|---|---|
| SIGNATURE OF PARENT/GUARDIAN | DATE |
| PRINTED NAME OF PARENT/GUARDIAN | |
| SIGNATURE OF PARENT/GUARDIAN Signature of Other Parent (Optional, unless required by the IRB.) | DATE |
| PRINTED NAME OF PARENT/GUARDIAN | |
| The IRB has determined that the signature of both parents is requ | ıired. |
| If not obtaining both parental signatures, please indicate reason below: | : |
| Other parent is deceased, unknown, incompetent, or not reasonal | bly available. |
| Parent/Guardian signing above has sole legal responsibility for the custody of the child. | e care and |
| The IRB has determined that the signature of both parents is No. | OT required. |
| ASSENT OF MINOR (Entire section must be completed if the participant's intellectual and less than 18 years. Participants with an intellectual age of 7 - required to sign.) | |
| If written assent is not obtained on an age-appropriate participant, checonot: | ck reason why |
| 1.) The participant's intellectual age is less than seven. | |
| 2.) The participant dissented, but the participant's parent(s)/guard intervention(s) or procedure(s) involved in the research hold out the podirect benefit that is important to the health and/or well being of the paravailable only in the context of this research study 3.) Other: | ssibility of a |

I have read and understand the description of this research. I have had a chance to

Protocol 2021-1059 NCT05360160 January 28, 2025 

I have been told what I will be asked to do in this study.

I have been told that I do not have to be in this study. If I decide not to be in this study, no one will be mad at me. I may quit at any time, but if I do, I may need to take a different treatment.

I have had a chance to talk about the study and ask the study doctor questions. All of my questions have been answered. I agree to be in this study and do what I am asked to do so long as I want to stay in this study. I agree that the study doctor can put me on this study. By signing this paper, I am not giving up any of my legal rights. I have been given a copy of this document.

| SIGNATURE OF MINOR (Age 13-17) | DATE |
|--------------------------------|------|
| PRINTED NAME OF MINOR | |